CLINICAL TRIAL: NCT01117220
Title: Four Week, Double Blind, Placebo Controlled Phase III Trial Evaluating The Efficacy, Safety And Pharmacokinetics Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
Brief Title: Safety And Efficacy Of Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed) (Protocol A1281196)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1281196
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder
Keywords: pediatric; bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Active Comparator)
  Interventions: Drug: Ziprasidone Oral Capsules

INTERVENTIONS:
Drug: Placebo — Placebo matching the oral ziprasidone capsules of 20,40, 60 and 80 mg in strength. Subjects will be dosed for 4 weeks using a flexible dose design with minimal dose range of 40 mg twice a day (BID) to maximum dose range of 80 mg BID (weight specific- < 45kg max dose 40 mg BID).
  Arms: 2
Drug: Ziprasidone Oral Capsules — Oral ziprasidone capsules of 20,40, 60 and 80 mg in strength. Subjects will be dosed for 4 weeks using a flexible dose design with minimal dose range of 40 mg twice a day (BID to maximum dose range of 80 mg BID (weight specific- < 45kg max dose 40 mg BID).
  Other Names: Geodon, Zeldox
  Arms: 1

SUMMARY:
The purpose of this study is to determine if flexibly-dosed ziprasidone is safe and effective for the treatment of children and adolescents (ages 10-17) with Bipolar l Disorder (Manic or Mixed).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria for Bipolar I disorder (manic or mixed)
* At the screening and baseline visits, subjects must have a Young Mania Rating Scale (YMRS) score of at least 17.
* The subject must have a Body Mass Index (BMI) z score between -1.65 and +2.00, inclusive

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator
* Any history of serious or unstable illness
* Risk for prolonged QT

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 4 in Young Mania Rating Scale (YMRS) total score. | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression of Severity (CGI S) score. | 4 weeks
Clinical Global Impression of Improvement (CGI I) score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281196&StudyName=Safety%20And%20Efficacy%20Of%20Ziprasidone%20In%20Children%20And%20Adolescents%20With%20Bipolar%20I%20Disorder%20%28Manic%20Or%20Mixed%29%20%28Protocol%20A1281196%29